CLINICAL TRIAL: NCT05053854
Title: Phase 1 Trial of PARP Inhibitor Combined With 177Lu-DOTA-Octreotate Peptide Receptor Radionuclide Therapy (PRRT) in Patients With Metastatic NeuroEndocrine Tumor
Brief Title: PARP Inhibitor With 177Lu-DOTA-Octreotate PRRT in Patients With Neuroendocrine Tumours
Acronym: PARLuNET
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMC67199
Record Dates: First submitted 2021-09-02; First posted 2021-09-23 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Neuroendocrine Tumors
Keywords: NET
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — talazoparib

STUDY DESIGN:
Intervention Model Description: Prospective single arm, single centre, Phase 1 study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 177Lu-DOTA-Octreotate + talazoparib (Experimental): Patients will receive 4 cycles of 177Lu-DOTA-Octreotate every 8 weeks, the last 3 cycles combined with talazoparib on days 2-6 of each cycle.
  Interventions: Drug: Talazoparib

INTERVENTIONS:
Drug: Talazoparib — During dose escalation, doses of talazoparib that can be administered are 0.1mg, 0.25mg, 0.5mg or 1mg oral daily. Talazoparib will be given on days 2-6 of each cycle of 177Lu-DOTA-Octreotate for cycles 2-4, every 8 weeks
  Other Names: Combination product: 177Lu-DOTA-Octreotate

SUMMARY:
This phase 1 dose-escalation study is designed to evaluate the safety and tolerability of talazoparib in combination with 177Lu-DOTA-Octreotate peptide receptor radionuclide therapy (PRRT) in patients with metastatic pancreatic or midgut neuroendocrine tumour (NET).

DETAILED DESCRIPTION:
This phase 1, single arm, single centre study is designed to evaluate the safety and tolerability of talazoparib in combination with 177Lu-DOTA-Octreotate in patients with metastatic NET.

Patients will receive 1 cycle of 177Lu-DOTA-Octreotate alone followed by 3 cycles of 177Lu-DOTA-Octreotate combined with 5 days of talazoparib.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be > or equal to18 years of age and must have provided written informed consent.
2. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
3. Histologically confirmed Grade 2 NET, Ki-67 of 3-20%, from pancreatic or intestinal origin.
4. Patient clinically suitable for PRRT
5. Tumor SSR uptake on GaTate PET/CT higher than liver activity, ≥ modified Krenning 3 score
6. No discordant FDG-avid disease on FDG PET/CT
7. No evidence of significant uncorrected carcinoid heart disease
8. Patients must be willing and able to comply with the protocol for the duration of the study including undergoing treatment, scheduled assessments
9. Patients must have adequate bone marrow, hepatic and renal function defined as:

   * Haemoglobin ≥100 g/L
   * Absolute neutrophil count ≥1.5x109/L
   * Platelets ≥150 x109/L
   * Total bilirubin ≤1.5 x upper limit of normal (ULN)
   * Aspartate transaminase (AST) (SGOT) and alanine transaminase (ALT) (SGPT)

     ≤2.5 x ULN if there is no evidence of liver metastasis or ≤5 x ULN in the presence of liver metastases.
   * Albumin ≥ 30 g/L
   * Adequate renal function: eGFR ≥ 50 ml/min

Exclusion Criteria:

1. Surgery or radiotherapy within <3 weeks of registration. Patients must have recovered from any effects of any major surgery.
2. Any prior exposure to peptide receptor radionuclide therapy (177Lu, 111In or 90Y labelled), PARPi, immunotherapy
3. Uncontrolled intercurrent illness that is likely to impede participation and /or compliance
4. Other malignancies unless curatively treated with no evidence of disease within previous 3-years other than adequately treated non-melanoma skin cancer or melanoma in situ.
5. Previous or current history of myelodysplastic syndrome/acute myeloid leukemia
6. Patients unable to swallow orally administered medications or with gastrointestinal disorders likely to interfere with the absorption of the study medication.
7. Use of strong P-gp inhibitors (eg, dronedarone, quinidine, ranolazine, verapamil, ketoconazole, itraconazole), P-gp inducers (eg, rifampin, tipranavir/ritonavir), or BCRP inhibitors (eg, elacridar [GF120918]) should be avoided.
8. Participation in another clinical study with an investigational product or another systemic therapy administered in the last 3 weeks (except short acting SSA).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-12-08 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose Talazoparib with 177Lu-DOTA-Octreotate | Through study completion, up to 18 months following first administration of PRRT.
  Maximum tolerated dose of Talazoparib when given in combination with 177Lu-DOTA-Octreotate
Dose limiting toxicity talazoparib | Each cohort of 3 patients be assessed for DLTs in the first 6 weeks (cycle 2) of treatment and a dose for the next cohort will be determined (each cycle is 8 weeks)
  The toxicity (haematologic or non-haematologic) that prevents further administration of the trial talazoparib treatment at that dose level.

SECONDARY OUTCOMES:
Adverse Events and Serious Adverse Events measured using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 | Through Study completion, up to 18 months after the last patient commences treatment.
  Safety of the combination will be measured by AEs and SAEs
Radiographic progression free survival | Through study completion, up to 18 months following first administration of PRRT.
  The time from treatment initiation to the first date of progression on imaging or death due to any cause. Imaging progression will be assessed by RECIST 1.1. Patients who commence new systemic therapy before evidence of disease progression on conventional imaging will be considered to have progressed.
Overall Survival | Through study completion, up to 18 months following first administration of PRRT.
  The time from treatment initiation to the date of death due to any cause. For patients alive, the time will be censored at the last time the patients was known to be alive.
Treatment discontinuation due to toxicity | Through study completion, up to 18 months following first administration of PRRT.
  The number of patients who discontinue treatment at any time due to treatment related toxicity will be reported and will be also categorised by dose level.
Rate of Treatment discontinuation due to toxicity | Through study completion, up to 18 months following first administration of PRRT.
  The percentage of patients who discontinue treatment due to treatment related toxicity will be reported and will be also categorised by dose level

CONTACTS AND LOCATIONS:
Locations (1):
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No